CLINICAL TRIAL: NCT04659850
Title: Do Dietary AGEs Have an Acute Effect on Metabolism and Cognition
Brief Title: Impact of AGEs on Metabolism & Cognition
Acronym: AGEs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2017/RI/5
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: No Conditions
MeSH Terms: interventions — Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: Dietary Challenge
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Group 1 participants in the young 18 - 30 age group
  Interventions: Other: low fat, low AGE milkshake; Other: low fat, high AGE milkshake; Other: high fat, low AGE; Other: high fat, high AGE milkshake
- Group 2 (Other): Group 2 participants in the older 55 - 75 age group
  Interventions: Other: low fat, low AGE milkshake; Other: low fat, high AGE milkshake; Other: high fat, low AGE; Other: high fat, high AGE milkshake

INTERVENTIONS:
Other: low fat, low AGE milkshake — low fat, low AGE milkshake given after an overnight fast
Other: low fat, high AGE milkshake — low fat, high AGE milkshake given after an overnight fast
Other: high fat, low AGE — high fat, low AGE milkshake given after an overnight fast
Other: high fat, high AGE milkshake — high fat, high AGE milkshake given after an overnight fast

SUMMARY:
A number of processed foods particularly those high in protein and based on whey protein are high in advanced glycation end products (AGEs). AGEs are the result of a chemical reaction between mainly sugar and protein when they are heated together (known as the Maillard reaction). Whey protein is routinely derived via high temperature processing methods which produce AGEs. AGEs are absorbed during digestion and high circulating concentrations of AGEs are associated with adverse health effects such as dementia and the metabolic syndrome. In this study we aim to firstly ascertain the habitual level of AGE intake in the diet via a dietary questionnaire and equate this to both metabolic health and cognition at baseline. Volunteers will then be given a milkshake with either a high or low AGE content on either a high or low fat background. AGEs are usually ingested as part of a processed food diet which can be high in fat and it is necessary to separate the effects of these two food types. We will test these effects in a young and older group of volunteers with low and higher levels of circulating AGEs respectively. Circulating levels of hormones, glucose and lipids in the blood will be measured as indicators of metabolic health. Cognitive tests will be carried out to assess the impact of AGEs on episodic memory.

DETAILED DESCRIPTION:
This study will be a short-term, randomized, double-blind, cross-over trial. Volunteers will be younger (18-30 years) and older (55-75 years) men and women, normal and overweight (BMI>19 to 29.9). N=24 in each age group.

Medical screening for all study volunteers and neuropsychological screening will be carried out prior to study start. A small, pin prick, fasted blood sample will be taken to measure glucose and HbA1C levels to rule out type 2 diabetics. Anthropometric and body composition measurements will also be taken. Body weight and height will be measured using a scale and a stadiometer to the nearest 0.5 kg and 0.5 cm, respectively. Waist and hip circumferences will be measured and the waist-to-hip ratio calculated. Standard procedures will be followed for the anthropometric measurements and the average of three measurements taken. Neuropsychological screening may be repeated on another day if volunteers are borderline on their first visit as scores may vary by a couple of points depending on external events i.e. vounteers are having a bad day. Experienced staff will carry out abdominal fat measurements by manual determination of the area between the upper surface of the second lumbar vertebra, the lower surface of the fourth lumbar vertebra, and the lateral margins of the outer rib cage. If the Viscan is available we will use that to measure abdominal fat. Venous blood samples will be collected as appropriate for the hormones and metabolites to be tested and stored at -70 °C.

The day prior to the challenge volunteers will visit the Human Nutrition Unit (HNU, RINH). They will be given a low AGE breakfast and be supplied with a low AGE lunch and dinner for that day and instructed not to consume anything else. After an overnight fast volunteers will receive a one-off dose of either high AGE (11.4 mgs) or low AGE (2.4 mgs) whey protein delivered in a either a low or high fat milkshake (400ml) blended with flavours and a consistent quantity of sugar. All ingredients will be commercially available and of food grade. Apart from differences in fat and AGE the content of shakes will be closely balanced for sugar and other components. All participants will be asked to answer two questionnaires one to determine their habitual intake of dietary AGEs and one to determine their level of physical activity.

The different milkshakes will be tested with a minimum 7 day wash out period between tests. Volunteers will be randomised to each test group. After a 12 h overnight fast and a standardised intake the day prior to the tests, and no strenuous physical activity for 2 days previously, subjects will attend the HNU. Volunteers will be requested to provide a small urine sample for AGE analysis. An intravenous catheter will then be placed in an antecubital vein and flushed with saline between aspirations to keep the catheter clear. After a short resting period, a blood sample will be taken prior to the first memory test then a single milkshake will be consumed under supervision. Blood samples will be taken immediately before the milkshake ingestion (0 min) and after 30, 60, 90, 120, 150 and 180 and 240 min. Further computer based memory tests will be carried out at 30, 90 and 240 minutes. A urine sample will be requested at the end of the study before participants are offered lunch. Memory tests have been designed by Dr Ros Langston (University of Dundee) and Dr Kevin Allan, School of Psychology and will be carried out on lap tops specifically designated for this study. Blood and urine will be analysed for AGEs. Blood will also be analysed for glucose lipids and hormones. Dr Janice Drew will also analyse blood samples for gene expression of the SIRT-1/NAD+ complex indicative of the response of individuals to dietary challenge.

ELIGIBILITY:
Inclusion Criteria:

* Heathy
* Sedentary
* 18-30 or
* 55-75

Exclusion Criteria:

* diagnosed type 2 diabetes,
* CVD
* history of neurological abnormalities
* current psycho-active medication
* current anti-inflammatory medication
* Current glucose lowering medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Impact of Advanced Glycation End Products on Metabolism and Cognition | Four weeks per participant
  Habitual AGE intake, determined from dietary questionnaires, specifically designed for this purpose, taken at the start of the study, will be correlated with levels of circulating AGEs and outcomes such as inflammatory markers and expression of genes associated with susceptibility to metabolic disease and acute response to dietary challenge will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Campbell, PHD, Principal Investigator — UoA Rowett Institute of Nutrition and Health
Locations (1):
- University of Aberdeen Rowett Institute of Nutrition and Health, Aberdeen, Scotland, United Kingdom